CLINICAL TRIAL: NCT03382795
Title: Retreatment With 1st Generation EGFR TKIs in Sensitizing EGFR Mutation Positive Non-Squamous Cell Carcinoma Patients Who Previously Treated With EGFR TKI and Cytotoxic Chemotherapy
Brief Title: Retreatment With Epidermal Growth Factor Receptor(EGFR) Tyrosine Kinase Inhibitor in EGFR Mutation Positive Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Chong Kun Dang Pharmaceutical Corp. (Industry)
Responsible Party: Principal Investigator, Sung Yong Lee, Professor, Korea University Guro Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MLCSG2017001
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: EGFR Positive Non-small Cell Lung Cancer
Keywords: Epidermal growth factor receptor tyrosine kinase inhibitor; Cytotoxic chemotherapy; Epidermal growth factor receptor mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EGFR retreat group (Experimental)
  Interventions: Drug: EGFR

INTERVENTIONS:
Drug: EGFR — Gefitinib 250mg or Erlotinib 150mg medication, Once-Daily.

SUMMARY:
In this trial, treatment efficacy and safety of retreatment with 1st generation epidermal growth factor receptor(EGFR) tyrosine kinase inhibitor(TKI)s(Gefitinib/Erlotinib), will be assessed in patients with sensitizing EGFR mutation positive Non-Squamous Cell Carcinoma patients who previously treated with EGFR TKI and cytotoxic chemotherapy

DETAILED DESCRIPTION:
This study is designed to be multi-center, open-label, single-arm, prospective, phase II trial of patient with sensitizing EGFR mutation positive Non-Squamous Cell Carcinoma patients who previously treated with EGFR TKI and cytotoxic chemotherapy. Approximately 69 patients will be enrolled into the trial, and expected study duration is 48 months from Institutional Review Board(IRB) and Korea Ministry of Food and Drug Safety(MFDS) approval date.

The study drug will be administered orally as one tablet(Gefitinib 250mg/ Erlotinib 150mg) once a day until disease progression or manifestation of unacceptable toxicity. The initial dose of the study drug daily can be reduced according to dose reduction criteria in protocol. A cycle of study treatment is defined as 28 days, and subjects will visit the site every 2 cycles(56 days).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 19 years of age
2. Non Small Cell Lung Cancer(Non-Squamous Cell Carcinoma) patients who had shown clinical benefits (Complete response(CR) or Partial response(PR) or Stable disease(SD) ≥6 months) from EGFR-TKIs as first line treatment and developed progressive disease, and then received cytotoxic chemotherapy more than 4 cycles and developed progressive disease, and then confirmed T790 negative and sensitizing EGFR mutation(E19Del, L858R, L861Q, G719X, E19insertion) positive in Histologic, cytologic specimen or blood.
3. Patient with at least one measurable lesions according to RECIST v 1.1
4. Expected life expectancy ≥ 12 weeks
5. Eastern Cooperative Oncology Group(ECOG) performance status ≤ 2
6. Patients who have proper hematologic, renal and hepatic functions as follows:

   * Absolute neutrophil count(ANC) ≥ 1,500/mm³
   * platelets ≥ 100,000/mm³
   * Hemoglobin ≥ 9g/dL
   * Total bilirubin ≤ 1.25 X UNL
   * Aspartate aminotransferase(AST or SGOT) and alanine aminotransferase(ALT or SGPT) ≤ 3.0 X UNL (if liver metastasis ≤5.0 X UNL)
   * Alkaline phosphatase ≤ 2.5 X UNL (if liver metastasis ≤5.0 X UNL)
   * Serum creatinine ≤ 1.5mg/dL
7. patients who are willing to comply with study procedure and voluntarily provide informed consent with signature

Exclusion Criteria:

1. Patients who have preexisting or coexisting malignancies in other parts except for effectively treated non-melanoma skin cancer, cervical carcinoma in situ(CIS) cervical cancer within the last 5 years
2. Patients with brain metastasis except for the followings:

   - Asymptomatic and stable brain metastases for which local treatment has been given: corticosteroids treatment isn't requiured for at least 2 weeks before starting the study treatment.
3. Patients currently receiving palliative radiation therapy or have toxicities from radiation therapy at screening.
4. Patients with clinically active history of interstitial lung disease(ILD), Drug induced ILD, Radiation pneumonitis
5. Patients with clinically significant cardiovascular disease or myocardial infarction within the past 12 months.
6. Patients with active infection or severe systemic disease that are difficult to include in this study
7. Patients who received radiation therapy to target lesion of this study.
8. Patients who had major operation within 4 weeks before starting the study treatment and were not fully recovered.
9. Patients who were administered other study drugs within 4 weeks before starting the study treatment
10. Males and females of reproductive potential who are not using an effective method of birth control and females who are pregnant or breastfeeding or have a positive pregnancy test prior to study entry
11. Patients who are difficult to include in this study in accordance with the investigator's judgment
12. Patients with histories of hypersensitivity to investigational product(IP) or any components of the agent
13. Patients with any of the following genetic predispositions including galactose intolerance, Lapp lactase deficiency, lactose intolerance or glucose-galactose malabsorption
14. Patient previously received cytotoxic chemotherapy within 2 weeks of IP administration
15. Patient received Immunotherapy prior to the study participation
16. Patients who are difficult to include in this study in accordance with the investigator's judgment due to severe adverse effects during previous EGFR TKI treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) including rage of CR&PR | Through study completion (5 years)
  Assessed on based of RECIST 1.1.

SECONDARY OUTCOMES:
Progression Free Survival, PFS | Through study completion (5 years)
  Progression-free survival (PFS) the time from first dose of the study drug until the date of disease progression or death by any cause
Overall Survival | Through study completion (5 years)
  Overall Survival (OR) the time from first dose of the study drug until the date of death by any cause
The incidence of Adverse Events(including Serious Adverse Events and Adverse Drug Reactions) | Through study completion (5 years)
  Assessment on the base of NCI-CTCAE (version 4.03)

CONTACTS AND LOCATIONS:
Overall Officials: Sung Yong Lee, MD, Ph.D., Principal Investigator — Professor
Locations (8):
- South Korea (8):
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Chungnam National University Hospital, Daejeon
  - Yonsei University Severance Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul

REFERENCES:
- [Background] Janssen-Heijnen ML, Coebergh JW. The changing epidemiology of lung cancer in Europe. Lung Cancer. 2003 Sep;41(3):245-58. doi: 10.1016/s0169-5002(03)00230-7. PMID 12928116
- [Background] Jemal A, Chu KC, Tarone RE. Recent trends in lung cancer mortality in the United States. J Natl Cancer Inst. 2001 Feb 21;93(4):277-83. doi: 10.1093/jnci/93.4.277. PMID 11181774
- [Background] Kinoshita FL, Ito Y, Nakayama T. Trends in Lung Cancer Incidence Rates by Histological Type in 1975-2008: A Population-Based Study in Osaka, Japan. J Epidemiol. 2016 Nov 5;26(11):579-586. doi: 10.2188/jea.JE20150257. Epub 2016 Apr 30. PMID 27150013
- [Background] Dela Cruz CS, Tanoue LT, Matthay RA. Lung cancer: epidemiology, etiology, and prevention. Clin Chest Med. 2011 Dec;32(4):605-44. doi: 10.1016/j.ccm.2011.09.001. PMID 22054876
- [Background] Shin A, Oh CM, Kim BW, Woo H, Won YJ, Lee JS. Lung Cancer Epidemiology in Korea. Cancer Res Treat. 2017 Jul;49(3):616-626. doi: 10.4143/crt.2016.178. Epub 2016 Sep 23. PMID 27669705
- [Background] Jackman DM, Miller VA, Cioffredi LA, Yeap BY, Janne PA, Riely GJ, Ruiz MG, Giaccone G, Sequist LV, Johnson BE. Impact of epidermal growth factor receptor and KRAS mutations on clinical outcomes in previously untreated non-small cell lung cancer patients: results of an online tumor registry of clinical trials. Clin Cancer Res. 2009 Aug 15;15(16):5267-73. doi: 10.1158/1078-0432.CCR-09-0888. Epub 2009 Aug 11. PMID 19671843
- [Background] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Background] Maemondo M, Inoue A, Kobayashi K, Sugawara S, Oizumi S, Isobe H, Gemma A, Harada M, Yoshizawa H, Kinoshita I, Fujita Y, Okinaga S, Hirano H, Yoshimori K, Harada T, Ogura T, Ando M, Miyazawa H, Tanaka T, Saijo Y, Hagiwara K, Morita S, Nukiwa T; North-East Japan Study Group. Gefitinib or chemotherapy for non-small-cell lung cancer with mutated EGFR. N Engl J Med. 2010 Jun 24;362(25):2380-8. doi: 10.1056/NEJMoa0909530. PMID 20573926
- [Background] Rosell R, Carcereny E, Gervais R, Vergnenegre A, Massuti B, Felip E, Palmero R, Garcia-Gomez R, Pallares C, Sanchez JM, Porta R, Cobo M, Garrido P, Longo F, Moran T, Insa A, De Marinis F, Corre R, Bover I, Illiano A, Dansin E, de Castro J, Milella M, Reguart N, Altavilla G, Jimenez U, Provencio M, Moreno MA, Terrasa J, Munoz-Langa J, Valdivia J, Isla D, Domine M, Molinier O, Mazieres J, Baize N, Garcia-Campelo R, Robinet G, Rodriguez-Abreu D, Lopez-Vivanco G, Gebbia V, Ferrera-Delgado L, Bombaron P, Bernabe R, Bearz A, Artal A, Cortesi E, Rolfo C, Sanchez-Ronco M, Drozdowskyj A, Queralt C, de Aguirre I, Ramirez JL, Sanchez JJ, Molina MA, Taron M, Paz-Ares L; Spanish Lung Cancer Group in collaboration with Groupe Francais de Pneumo-Cancerologie and Associazione Italiana Oncologia Toracica. Erlotinib versus standard chemotherapy as first-line treatment for European patients with advanced EGFR mutation-positive non-small-cell lung cancer (EURTAC): a multicentre, open-label, randomised phase 3 trial. Lancet Oncol. 2012 Mar;13(3):239-46. doi: 10.1016/S1470-2045(11)70393-X. Epub 2012 Jan 26. PMID 22285168
- [Background] Sequist LV, Yang JC, Yamamoto N, O'Byrne K, Hirsh V, Mok T, Geater SL, Orlov S, Tsai CM, Boyer M, Su WC, Bennouna J, Kato T, Gorbunova V, Lee KH, Shah R, Massey D, Zazulina V, Shahidi M, Schuler M. Phase III study of afatinib or cisplatin plus pemetrexed in patients with metastatic lung adenocarcinoma with EGFR mutations. J Clin Oncol. 2013 Sep 20;31(27):3327-34. doi: 10.1200/JCO.2012.44.2806. Epub 2013 Jul 1. PMID 23816960
- [Background] Yu HA, Arcila ME, Rekhtman N, Sima CS, Zakowski MF, Pao W, Kris MG, Miller VA, Ladanyi M, Riely GJ. Analysis of tumor specimens at the time of acquired resistance to EGFR-TKI therapy in 155 patients with EGFR-mutant lung cancers. Clin Cancer Res. 2013 Apr 15;19(8):2240-7. doi: 10.1158/1078-0432.CCR-12-2246. Epub 2013 Mar 7. PMID 23470965
- [Background] Besse B, Adjei A, Baas P, Meldgaard P, Nicolson M, Paz-Ares L, Reck M, Smit EF, Syrigos K, Stahel R, Felip E, Peters S; Panel Members; ESMO. 2nd ESMO Consensus Conference on Lung Cancer: non-small-cell lung cancer first-line/second and further lines of treatment in advanced disease. Ann Oncol. 2014 Aug;25(8):1475-84. doi: 10.1093/annonc/mdu123. Epub 2014 Mar 25. PMID 24669016
- [Background] Asahina H, Oizumi S, Inoue A, Kinoshita I, Ishida T, Fujita Y, Sukoh N, Harada M, Maemondo M, Saijo Y, Dosaka-Akita H, Isobe H, Nukiwa T, Nishimura M; Hokkaido Lung Cancer Clinical Study Group. Phase II study of gefitinib readministration in patients with advanced non-small cell lung cancer and previous response to gefitinib. Oncology. 2010;79(5-6):423-9. doi: 10.1159/000326488. Epub 2011 Apr 8. PMID 21474967
- [Background] Koizumi T, Agatsuma T, Ikegami K, Suzuki T, Kobayashi T, Kanda S, Yoshikawa S, Kubo K, Shiina T, Takasuna K, Matsuo A, Hayasaka M, Morikawa M, Ameshima S. Prospective study of gefitinib readministration after chemotherapy in patients with advanced non-small-cell lung cancer who previously responded to gefitinib. Clin Lung Cancer. 2012 Nov;13(6):458-63. doi: 10.1016/j.cllc.2012.01.006. Epub 2012 Mar 7. PMID 22402083
- [Background] Oh IJ, Ban HJ, Kim KS, Kim YC. Retreatment of gefitinib in patients with non-small-cell lung cancer who previously controlled to gefitinib: a single-arm, open-label, phase II study. Lung Cancer. 2012 Jul;77(1):121-7. doi: 10.1016/j.lungcan.2012.01.012. Epub 2012 Feb 12. PMID 22333554
- [Background] Hata A, Katakami N, Yoshioka H, Fujita S, Kunimasa K, Nanjo S, Otsuka K, Kaji R, Tomii K, Iwasaku M, Nishiyama A, Hayashi H, Morita S, Ishida T. Erlotinib after gefitinib failure in relapsed non-small cell lung cancer: clinical benefit with optimal patient selection. Lung Cancer. 2011 Nov;74(2):268-73. doi: 10.1016/j.lungcan.2011.03.010. Epub 2011 May 6. PMID 21529987
- [Background] Kaira K, Naito T, Takahashi T, Ayabe E, Shimoyama R, Kaira R, Ono A, Igawa S, Shukuya T, Murakami H, Tsuya A, Nakamura Y, Endo M, Yamamoto N. Pooled analysis of the reports of erlotinib after failure of gefitinib for non-small cell lung cancer. Lung Cancer. 2010 Apr;68(1):99-104. doi: 10.1016/j.lungcan.2009.05.006. Epub 2009 Jun 21. PMID 19540616
- [Background] Mok TS, Wu Y-L, Ahn M-J, Garassino MC, Kim HR, Ramalingam SS, Shepherd FA, He Y, Akamatsu H, Theelen WS, Lee CK, Sebastian M, Templeton A, Mann H, Marotti M, Ghiorghiu S, Papadimitrakopoulou VA; AURA3 Investigators. Osimertinib or Platinum-Pemetrexed in EGFR T790M-Positive Lung Cancer. N Engl J Med. 2017 Feb 16;376(7):629-640. doi: 10.1056/NEJMoa1612674. Epub 2016 Dec 6. PMID 27959700
- See also: GLOBOCAN 2012: estimated cancer incidence, mortality and prevalence worldwide in 2012. All cancers (excluding nonmelanoma skin cancer) estimated incidence, mortality and prevalence worldwide in 2012 [Internet]. Geneva: World Health Organization — http://globocan.iarc.fr